CLINICAL TRIAL: NCT01582438
Title: A Local, Multicentre, Open Label Access Study, To Provide Sildenafil Therapy For Subjects Who Completed A1481156 Study And Are Judged By The Investigator To Derive Clinical Benefit From Continued Treatment With Sildenafil For Subjects In India
Brief Title: An Open Label Access Study For Subjects Who Completed A1481156
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481304
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Access program - sildenafil citrate, Viagra, Revatio — The recommended dose is 20 mg TID for subjects with body weight > 20 kg and 10 mg TID for subjects with body weight ≤ 20 kg. If subject is 18 years of age or older, the recommended dose is 20 mg TID, regardless of body weight. If a subject was receiving a higher dose in study A1481156 and the investigator believes that the subject requires continued treatment on that dose, or if dose reduction is judged to be associated with pulmonary arterial hypertension (PAH) deterioration in a particular subject, the higher dose may be made available, as judged on an individual basis on discussion with the sponsor.
  Other Names: sildenafil citrate, Viagra, Revatio

SUMMARY:
The purpose of this study is to provide sildenafil therapy to subjects who have completed the A1481156 study for the treatment of Pulmonary Arterial Hypertension (PAH) in India and are judged by the Investigator to derive clinical benefit from continued treatment with sildenafil citrate. Sildenafil citrate will be supplied for the treatment of Pulmonary Arterial Hypertension (PAH) until the subject continues to derive benefits from the treatment. The treating physicians (and the sponsor) will be responsible for reporting serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed study A1481156 and are judged by the Investigator to derive clinical benefit from continuous treatment with sildenafil citrate therapy.
* Subjects with pulmonary arterial hypertension (PAH ) being treated at a study site in India
* Subjects who are willing and able to comply with scheduled visits, treatment plan, and other study procedures

Exclusion Criteria:

* Pregnant or lactating female subjects.
* Current participation in other studies and during study participation, except for the A1481304 follow-up period.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- CARE Hospital, Hyderabad, Andhra Pradesh, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481304&StudyName=An%20Open%20Label%20Access%20Study%20For%20Subjects%20Who%20Completed%20A1481156